CLINICAL TRIAL: NCT07220174
Title: Pilot Usability Evaluation of GI Genius™ XR Software Running on a Virtual Reality Headset During Routine CRC Screening and Surveillance Colonoscopies
Brief Title: Use of GI Genius™ XR Software in Virtual Reality Headset During Routine Colonoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmo Artificial Intelligence-AI Ltd (Industry)
Responsible Party: Sponsor
Organization: Cosmo Pharmaceuticals NV (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CB-30-08/01
Record Dates: First submitted 2025-10-09; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Colonoscopy (Procedure)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Endoscopist with software GI Genius™ XR in headset (Experimental)
  Interventions: Device: software GI Genius™ XR on headset

INTERVENTIONS:
Device: software GI Genius™ XR on headset — The screening or surveillance colonoscopy is performed with the endoscopist wearing the headset and using the software GI Genius™ XR.

SUMMARY:
This pilot study will evaluate the usability and safety of software GI Genius™ XR in the Apple Vision Pro™ virtual reality headset when used in conjunction with the GI Genius™ system during routine screening and surveillance colonoscopy procedures. GI Genius™ XR enables colonoscopists to view the standard live endoscopic video feed within a virtual reality environment as an alternative to the conventional endoscopy tower display. The system provides a virtual screen that mirrors the tower video output without any image analysis or interpretation, allowing users to adjust screen size and position for optimal visualization and situational awareness.

ELIGIBILITY:
Inclusion Criteria for patient:

* Male or female aged ≥ 45 years;
* Scheduled for routine CRC screening or surveillance colonoscopy;
* Written informed consent to participate.

Inclusion Criteria for endoscopist:

* Male or female board-certified gastroenterologists experienced with CRC screening and surveillance colonoscopy;
* Written informed consent to participate.

Exclusion Criteria for patient:

* Not able to comply with the protocol requirement;
* Implanted or worn medical device (pacemaker, defibrillator, insulin pump, etc.).

Exclusion Criteria for endoscopist:

* Not able to comply with the protocol requirement;
* Implanted or worn medical device (pacemaker, defibrillator, insulin pump, etc.);
* Risk of falls;
* Seizures;
* Heart disease;
* Pregnant;
* Migraines;
* Eye or vision disorder;
* Inner ear disorder;
* Psychological disorder.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Day 1
  Collection and analysis of any adverse event.
GI Genius™ XR critical tasks | Day 1
  Correct execution of critical tasks through a questionnaire
Use effects | Day 1
  Use effects of the virtual reality headset on endoscopists through a questionnaire.
Problem resolution process | Day 1
  Management of non-specific problem resolution through a questionnaire.
Time management | During the procedure
  Time to complete key tasks during the procedure.
Interruption management | Day 1
  Number and severity of interruptions related to headset messages or other user device interactions.
User feedback on usability | Day 1
  Thematic analysis of qualitative feedback on headset integration.

SECONDARY OUTCOMES:
System Usability Score | Through study completion, an average of 3 months
  System Usability Score questionnaire across all participating endoscopists on a [0-100] scale, where 100 is the maximum positive outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States